CLINICAL TRIAL: NCT00451386
Title: A Prospective, Multicenter, Double-Blind, Randomized, Comparative Study to Evaluate the Safety, Local Tolerability, and Clinical Outcome of Ertapenem Versus Ceftriaxone in Pediatric Patients With Complicated Urinary Tract Infection, Skin and Soft Tissue Infection, or Community-Acquired Pneumonia
Brief Title: Ertapenem Study in Pediatric Patients Who Have Urinary Tract Infections, Skin Infections or Community-acquired Pneumonia (0826-036)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0826-036; 2007_525
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Urinary Tract Infections; Bacterial Pneumonia; Soft Tissue Infections
MeSH Terms: conditions — Urinary Tract Infections; Pneumonia, Bacterial; Soft Tissue Infections | interventions — Ertapenem; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0826, ertapenem sodium /Duration of Treatment: 14 Days
Drug: Comparator: ceftriaxone sodium /Duration of Treatment: 14 Days

SUMMARY:
This study will investigate the safety and efficacy of ertapenem versus ceftriaxone in pediatric patients with urinary tract infections, skin infections, or community-acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with UTI must have white blood cells and bacteria in the urine with bladder catheterization or urologic abnormality, kidney infection or both
* Patients with SSTI must have a recent infection
* Patients with CAP must have a chest x-ray indicating bacterial pneumonia and a fever

Exclusion Criteria:

* Patients with complete urinary tract blockage or kidney abscess
* Patients with infected burn wounds, bone infection, or bacterial arthritis
* Patients on mechanical ventilation or those with cystic fibrosis, chronic lung disease or puss in the space between the chest wall and lung

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400
Dates: Start 2002-01; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the incidence of any clinical and/or laboratory drug-related serious adverse experience during the parenteral therapy period in pediatric patients treated with ertapenem.

SECONDARY OUTCOMES:
To compare the safety of ertapenem versus ceftriaxone during the parenteral therapy period with respect to the proportion of patients with any drug-related adverse experiences in pediatric patients with UTI, SSTI, or CAP.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Arguedas A, Cespedes J, Botet FA, Blumer J, Yogev R, Gesser R, Wang J, West J, Snyder T, Wimmer W; Protocol 036 Study Group. Safety and tolerability of ertapenem versus ceftriaxone in a double-blind study performed in children with complicated urinary tract infection, community-acquired pneumonia or skin and soft-tissue infection. Int J Antimicrob Agents. 2009 Feb;33(2):163-7. doi: 10.1016/j.ijantimicag.2008.08.005. Epub 2008 Oct 21. PMID 18945594
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html